CLINICAL TRIAL: NCT06400407
Title: Lesion Network Mapping Navigated Continuous Theta-burst Stimulation for Motor Recovery in Acute Ischemic Stroke:A Randomized, Double-Blind, Sham-Controlled, Phase 2 Pilot Trial
Brief Title: Lesion Network MApping Navigated Continuous Theta-burst STimulation for Motor REcovery in Acute Ischemic Stroke
Acronym: MASTRE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HX-C-2024001
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Acute Ischemic
Keywords: Continuous Theta-burst Stimulation; Acute ischemic stroke; Motor recovery; Lesion network mapping; Navigation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To ensure the blind method, the sham stimulation coil will be used, which has the same parameters (including stimulation frequency, time, etc.) as the cTBS group, and has the same stimulation sound to ensure no effective stimulation, to ensure the blind state is maintained during the test. Investigators and patients who participate in the study treatment or are involved in the clinical evaluation of patients will be blinded to treatment grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Theta-burst Stimulation (Experimental): Based on the map, an 8-shaped coil was used to stimulate the motor function-related targets. The stimulation intensity was RMT80%, 600 pulses, 50Hz, 40s per target, and the stimulation interval was more than 2 hours. The treatment course lasted for 7 days.
  Interventions: Device: Continuous Theta-burst Stimulation
- Sham stimulation (Sham Comparator): A Sham stimulation coil was used to stimulate based on the map. The sound and duration were the same as the cTBS group, ensuring no effective stimulation. The treatment course lasted for 7 days.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Continuous Theta-burst Stimulation — Based on the map, an 8-shaped coil was used to stimulate the motor function-related targets. The stimulation intensity was RMT80%, 600 pulses, 50Hz, 40s per target, and the stimulation interval was more than 2 hours. The total course of treatment lasted 7 days.
  Arms: Continuous Theta-burst Stimulation
Device: Sham stimulation — A Sham stimulation coil was used to stimulate based on the map. The sound and duration were the same as the cTBS group, ensuring no effective stimulation. The total course of treatment lasted 7 days.
  Arms: Sham stimulation

SUMMARY:
This is a multicenter, sham-controlled, double-blind, randomized clinical trial to evaluate the efficacy and safety of lesion network mapping navigated cTBS in improving motor function in patients with acute ischemic stroke at 3-14 days after onset.

DETAILED DESCRIPTION:
The target population of this study was patients with acute ischemic stroke. Lesion network mapping and navigation were used to select individual stimulation targets. Enrolled patients were randomly assigned in a 1:1 ratio to the "cTBS group" or the "Sham stimulation group" and received:

cTBS group: Based on the map, an 8-shaped coil was used to stimulate the motor function-related targets. The stimulation intensity was RMT80%, 600 pulses, 50Hz, 40s per target, and the stimulation interval was more than 2 hours. The total course of treatment lasted 7 days.

Sham stimulation group: A Sham stimulation coil was used to stimulate based on the map. The sound and duration were the same as the cTBS group, ensuring no effective stimulation. The total course of treatment lasted 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old.
2. Acute ischemic stroke confirmed by CT or MRI at 3-14 days after onset.
3. Pre-stroke modified Rankin scale (mRS) score≤1.
4. 4≤NIHSS score≤ 25, 1a≤1, NIHSS5a/5b/6a/6b≥2 at least.
5. Moderate or severe motor dysfunction (Fugl-Meyer motor score < 80).
6. Written informed consent from patients or their legally authorized representatives.

Exclusion Criteria:

1. TMS contraindications include metallic foreign bodies in the head, pacemaker, implantable drug pumps, cochlear implants, etc.
2. Epilepsy or history of epilepsy, intracranial hypertension, tumor and other serious neurological disorders;
3. Midline displacement and brain parenchymal mass effect seen in head CT and other images;
4. Head CT or MRI showed bilateral acute cerebral infarction;
5. Evidence of acute intracranial hemorrhage;
6. A history of congenital or acquired hemorrhagic disease, coagulation factor deficiency, or thrombocytopenia disease;
7. After blood pressure control, the systolic blood pressure was still ≥180 mmHg or the diastolic blood pressure was ≥110 mmHg;
8. Patients during pregnancy or lactation and within 90 days of planned pregnancy;
9. Patients with severe mental disorders or dementia who can not cooperate with informed consent and follow-up;
10. Patients with malignancy or severe systemic disease and expected survival of less than 90 days;
11. Participants in other clinical intervention studies within 30 days before randomization or who were participating in other clinical intervention studies.
12. Patients with ataxia (NIHSS 7 ≥ 1) and aphasia (NIHSS 9 ≥ 2).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Improvement of motor function | 7 days
  Fugl-Meyer motor function score (FMMS) change from baseline at 7 days. FMMS 0-100 (higher score indicates better)
Serious adverse events ( SAEs ) | 7 days
  Serious adverse events ( SAEs )

SECONDARY OUTCOMES:
Early neurological improvement (ENI) | 7 days
  The proportion of patients with a reduction of ≥4 on the NIHSS, compared with the baseline score or an NIHSS of 0 or 1. NIHSS 0-42 (lower score indicates better)
Improvement of motor function | 90 days
  Fugl-Meyer motor function score (FMMS) change from baseline at 90 days. FMMS 0-100 (higher score indicates better)
Excellent functional outcome | 90 days
  Proportion of excellent functional outcome defined as an modified Rankin Scale (mRS) score ≤ 1 at 90 days. mRS 0-6 (lower score indicates better)
Barthel index of ADL | 90 days
  Barthel index of ADL, 0-100 (higher score indicates better)
EQ-5D-5L | 90 days
  he Health Questionnaire (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems."
Symptomatic intracranial hemorrhage | 7 days
  Proportion of symptomatic intracranial hemorrhage (sICH)
Symptomatic intracranial hemorrhage | 90 days
  Proportion of symptomatic intracranial hemorrhage (sICH)
Mortality | 90 days
  Rate of death from any cause within 90 days
Adverse events ( AEs ) | 90 days
  Rate of adverse events ( AEs ) within 90 days
Stroke recurrence | 90 days
  Cerebral infarction, cerebral hemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Ding L, Liu H, Jing J, Jiang Y, Meng X, Chen Y, Zhao X, Niu H, Liu T, Wang Y, Li Z. Lesion Network Mapping for Neurological Deficit in Acute Ischemic Stroke. Ann Neurol. 2023 Sep;94(3):572-584. doi: 10.1002/ana.26721. Epub 2023 Jun 27. PMID 37314250